CLINICAL TRIAL: NCT04121195
Title: A Phase 3, Open-label, Dose Escalation Study to Determine the Pharmacokinetics of Atazanavir Administered With RIfampicin to HIV Positive Adults on sEcond-line ART Regimen With Suppressed HIV-1 Viral Load (DERIVE)
Brief Title: Dose Escalation Study to Determine the Pharmacokinetics of Atazanavir Administered With RIfampicin to HIV Positive Adults on sEcond-line ART Regimen With Suppressed HIV-1 Viral Load
Acronym: DERIVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (Funder) (Unknown); Joint Clinical Research Centre, Kampala, Uganda (Unknown); University of Cape Town, Cape Town, South Africa (Unknown); Makerere University (Other); University of Turin, Turin, Italy (Unknown)
Responsible Party: Principal Investigator, Catriona Waitt, Chief Investigator, University of Liverpool
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DERIVE
Record Dates: First submitted 2019-10-02; First posted 2019-10-09 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: HIV/AIDS; Tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis

STUDY DESIGN:
Intervention Model Description: This is a dose-escalation study where pharmacokinetic assessments will be undertaken after dose-adjustments. In this type of study, each participant will serve as their own control, allowing the changes brought about by each dose change to be understood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation sequence (all participants) (Other): The trial will enrol virologically suppressed HIV infected volunteers who are stable on ATV/r and 2 NRTI containing ART following stringent screening to rule out evidence of renal, hepatic or gastrointestinal dysfunction which may affect the PK evaluation. A steady-state PK (PK1) sample collection shall be done on day 7 (+/-3) after enrolment. RIF will be added at standard dose (600 mg once daily) with a further PK evaluation 14 days later (PK2); due to the potential risk of sub therapeutic PI concentrations and emergence of HIV drug resistant strains, these individuals will be given DTG 50 mg twice daily for the duration of the dose-escalation study. ATV/r dose will be increased in a single step to the total modelled dose (PK3), given as twice daily doses. Once at maximum ATV/r dose, RIF will be increased to 1200 mg once a day for a further seven days (PK4). RIF will then be stopped, ATV/r stepped down to 300/100mg once a day and DTG continued for a further one week.
  Interventions: Drug: Dose escalation

INTERVENTIONS:
Drug: Dose escalation — The trial will enrol virologically suppressed HIV infected volunteers who are stable on ATV/r and 2 NRTI containing ART following stringent screening to rule out evidence of renal, hepatic or gastrointestinal dysfunction which may affect the PK evaluation. A steady-state PK (PK1) sample collection shall be done on day 7 (+/-3) after enrolment. RIF will be added at standard dose (600 mg once daily) with a further PK evaluation 14 days later (PK2); due to the potential risk of sub therapeutic PI concentrations and emergence of HIV drug resistant strains, these individuals will be given DTG 50 mg twice daily for the duration of the dose-escalation study. ATV/r dose will be increased in a single step to the total modelled dose (PK3), given as twice daily doses. Once at maximum ATV/r dose, RIF will be increased to 1200 mg once a day for a further seven days (PK4). RIF will then be stopped, ATV/r stepped down to 300/100mg once a day and DTG continued for a further one week.

SUMMARY:
The standard treatment for TB consists of rifampicin (RIF) as part of the regimen. However, due to drug-drug interactions (DDI), the bioavailability of PIs is greatly reduced when co-administered with RIF necessitating use of higher doses of the PI to overcome this effect. However, the potential effect of this increased dose on the DDI with bPIs is uncertain. Though some data has been collected that shows safe use of higher doses of LPV to overcome the DDI with standard doses of RIF in HIV-infected individuals, no substantive data has been collected on ATV to correctly adjust its dose when co-administered with RIF-based TB treatment.

Physiologically-based pharmacokinetic (PBPK) modelling was developed to understand ATV and RIF DDIs, and identified potential dosing strategies to overcome this challenge in adults and special populations under workpackage 1 of the VirTUAL consortium. From this work, it is anticipated that the dose of ATV/r should be increased from 300/100 once daily to 300/100mg twice daily in order to overcome the interaction with rifampicin and attain therapeutic plasma concentrations.

This dose escalation trial aims to:

1. Evaluate the steady state plasma and intracellular PK of ATV/r, when administered in adjusted (PBPK model-predicted) doses concurrently with RIF
2. Evaluate the safety and tolerability / acceptability of the adjusted dose of ATV/r that provides the therapeutic concentration when co-administered with RIF.
3. Evaluate the concentration of dolutegravir (DTG) and RIF when co-administered and explore the potential DDI with ATV/r

DETAILED DESCRIPTION:
Background and Justification

Both HIV and TB can successfully be managed using the currently available medications with the latter being curable. However, due to the detrimental drug-drug interaction (DDI) between RIF and the bPIs, there is a challenge in the management of the two conditions concurrently in persons who need both classes of drugs. RIF is a strong inducer of the hepatic enzyme cytochrome P450 (CYP) 34A which metabolizes several agents including the PI drugs thereby reducing their bioavailability. While rifabutin, an alternative rifamycin is associated with less DDI with bPI and maybe a better alternative to RIF in such circumstances, its cost, toxicity and lack of co-formulated preparations renders it to be a less likely sustainable option especially in LRS.

Though data published in 2008 showed a high incidence of adverse events when higher adjusted doses of LPV/r were used to overcome the DDI effect with RIF among healthy volunteers, data in 2012 among HIV-infected adults treated with adjusted doses of LPV/r co-administered with RIF-based TB treatment showed the drug was well tolerated with no significant adverse events. The major difference is that the 2012 study was conducted among HIV infected patients, that were already on normal doses of LPV/r and RIF at the time of enrolment who underwent PI dose escalation unlike the 2008 study among healthy volunteers who received the RIF and shortly after higher than normal doses of LPV/r in short succession with no step-wise phase to allow compensation. Similarly to LPV, ATV is affected by the inducing effect of RIF on the drug metabolizing enzyme cytochrome P450 (CYP) 34A, thereby significantly reducing its bioavailability to sub-therapeutic levels when co-administered in standard doses with RIF.

Several studies exploring the interaction between ATV/r and RIF have reached similar conclusions to the experience with LPV/r and RIF: A study in healthy volunteers given RIF first, then ATV/r first at standard dose with proposed dose escalation was halted when the first three participants developed hepatotoxicity. It was noted that the pre-induction of giving RIF first could have caused this problem. This argument is supported by a study conducted by Burger and colleagues where participants were first given ATV/r before the addition of RIF and where no hepatotoxicity occurred; in that study, the dose escalation evaluated was insufficient to overcome the interaction, but concluded that further evaluation was safe and appropriate. Similarly, Acosta and colleagues concluded that increased unboosted ATV was safe for co-administration with RIF, but that higher doses are required to overcome the DDI. No studies have yet evaluated this interaction in HIV-infected individuals.

It is notable that all of the currently available PIs have been associated with transient and usually asymptomatic elevations in serum aminotransferase levels, and ATV has been associated with mild-to-moderate elevations in indirect and total bilirubin concentration. All studied PIs are rare causes of clinically apparent, acute liver injury. The protease inhibitors are heterogeneous molecules with little structural similarity, most of which are peptide-like and resemble the short peptide that is cleaved by the viral protease; for this reason, the patterns of liver toxicity will differ between drugs of this class.

A recent study seeking to evaluate an increased dose of the bPI ritonavir boosted darunavir (DRV/r) in combination with rifampicin resulted in rates of hepatotoxicity which necessitated the trial to be halted on the advice of the IDSMB (CROI 2019 Abstract 81). These trial participants had been stable on treatment with LPV/r and were transitioned to DRV/r for the trial; the alteration in liver enzymes became apparent early on, and may have resulted in part from the change in bPI administered to the patient.

For the reasons detailed in the paragraphs above in consideration of the previous studies investigating either LPV/r, ATV/r or DRV/r in conjunction with RIF, we have chosen the study population of healthy HIV-infected patients who are already stable on treatment with standard dose of ATV/r, and who will have RIF introduced at a time when they will be at equilibrium as regards the ATV/r. Continuation on ATV/r at standard dose together with RIF for a two week period will enable a further equilibrium to have been established prior to escalation of the bPI dose. Both of these considerations may reduce the likelihood of hepatotoxicity, although frequent monitoring of safety bloods will be undertaken.

RIF also affects the bioavailability of DTG, however, this is effectively overcome by administering DTG twice daily as opposed to the standard once-a-day dose; the elevated dose of DTG has not been associated with concerns relating to liver toxicity.

As part of the VirTUAL consortium, physiologically-Based Pharmacokinetic (PBPK) modelling was done at the University of Liverpool to characterize bPI and RIF DDIs. Dosing strategies were identified / predicted to overcome the DDI between bPI and RIF that informed the ATV doses that shall be used in this trial to predict the most appropriate dose of ATV given with a standard dose RIF. From this work, it is predicted that increasing the dose of boosted ATV from ATV/r 300/100mg once daily to 300/100mg twice daily will achieve sufficient plasma concentrations when ATV/r is to be given in combination with RIF. The PBPK model utilised for this prediction was developed considering a mathematical description of the molecular and physiological processes underpinning the distribution of ATV/r and RIF. Experimental and clinical data were integrated into a computational framework developed using MATLAB and Simbiology and validated following international guidelines.

The RIF induction potential on Phase I enzyme and transporters expression, the RIF inhibitory effect on uptake transporters and the RTV inhibitory effect on CYP3A4 were all mathematically described for the simulation of the DDI. The PBPK model was qualified considering available clinical data for CYP3A4 probe (midazolam) and ATV ± RTV alone at different doses (400mg q.d unboosted, 300/100 mg q.d boosted) or in combination with RIF as previously described. The qualification was based on the calculation of the absolute average fold error (AAFE) and root mean squared error (RMSE) where appropriate. AAFE is a useful parameter to assess over or under-prediction of the model, values closer to 1 indicates a closer similarity with observed values. RMSE calculates the error between the predicted value and the observed value. RMSE is particularly sensitive to outliers and values closer to zero indicate a reliable prediction. The model was assumed to be qualified if the simulated values were within 2-fold of the mean reported values, AAFE <2 and RMSE <1 as per convention for the approach. Dose adjustment to overcome the effect of RIF on ATV/r was simulated considering available formulations with the overall of achieving ATV exposure comparable to established regimens (e.g. 300/100mg q.d) without RIF.

This study therefore aims to evaluate the steady state of the PBPK modelled adjusted doses of ATV given in different doses in HIV-1 infected adults on second line therapy with suppressed viral load so as to determine the most appropriate dose to be used concurrently with RIF. The study will evaluate baseline ATV/r concentrations in participants who have been treated with this agent for many months, then evaluate the impact of the addition of RIF, before evaluating ATV/r at the full modelled dose (300/100 twice daily) with a final step to consider the impact of increased doses of RIF (from standard dosing of 600 mg once daily to 1200 mg once daily).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide a signed and dated informed consent
2. HIV positive male or female ≥ 18 years of age
3. 50 - 75kg of weight
4. On ATV/rand 2 nucleos(t)ide reverse transcriptase inhibitor containing ART regimen for at least 6 months
5. Undetectable HIV viral load (<50 copies/ml) at screening PLUS an undetectable VL during the most recent test done between 6 and 12 months prior to screening.
6. A negative pregnancy test for females of child-bearing potential. Should also not be breast feeding.
7. On or willing to use effective contraception for at least 4 weeks prior to enrolment, throughout the study period and at least 4 weeks after end of the study(please see section 10.3 for a detailed definition of effective contraception for this study).
8. Clinically stable with no AIDS defining illness within the past 6 months.
9. A normal chest x-ray
10. Ability and willingness to understand and adhere to the study procedures for the entire study duration.
11. Able to attend for regular study follow-up visits

Exclusion Criteria:

1. Any clinical contraindications to the use of ATV/r, DTG or RIF.
2. Currently receiving treatment for tuberculosis
3. Hepatitis B surface antigen positive or Hepatitis C Antibody positive.
4. Requirement for concomitant medication with known major interactions with study drugs
5. Current participation in another clinical trial or research protocol
6. Symptoms of TB

   * weight loss > 2.5% in 4 weeks;
   * cough > 2 weeks;
   * night sweats> 2 weeks;
   * fever > 2 weeks;
7. Clinical or laboratory evidence of any of the following:

   * AST/ALT > 1.5 x the upper limit of normal range (ULN)
   * AST/ALT > 1.0 x ULN
   * > 125 mg/dl fasting serum glucose;
   * Serum creatinine ≥ 1.5 X ULN in the absence of dehydration. Or estimated glomerular filtration rate <60mL/min according to Cockcroft-Gault formula for creatinine clearance.
8. Moderate to severe anaemia (Haemoglobin level < 8 g/dL)
9. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study. The investigator should make this determination in consideration of the patient's medical history, clinical and/or laboratory results.
10. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
11. Known chronic underlying disease such as sickle cell disease, diabetes and severe cardiac impairment.
12. Inability to tolerate oral medication, or to drink.
13. Patients taking drugs that are strong inducers of CYP3A4 such as carbamazepine and phenytoin.
14. Known hypersensitivity to any of the agents used in the study
15. Patients with prior herbal medication within one week of screening
16. Use of other investigational drugs within 30 days of enrolment
17. Patients taking medications prohibited by the protocol (see appendix 5)
18. History of substantial use of alcohol that interferes with expected normal activities as determined by the investigator. Additionally, alcohol should be avoided throughout the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Plasma Cmax of ritonavir-boosted Atazanavir | 18 months
  The steady state plasma Cmax of ATV/r when administered in adjusted (PBPK model-predicted) doses (300/100mg twice daily) concurrently with standard dose of RIF (600mg) in HIV infected individuals.
Plasma AUC of ritonavir-boosted Atazanavir | 18 months
  The steady state plasma AUC of ATV/r when administered in adjusted (PBPK model-predicted) doses (300/100mg twice daily) concurrently with standard dose of RIF (600mg) in HIV infected individuals.
Plasma Clearance of ritonavir-boosted Atazanavir | 18 months
  The steady state plasma CL of ATV/r when administered in adjusted (PBPK model-predicted) doses (300/100mg twice daily) concurrently with standard dose of RIF (600mg) in HIV infected individuals.
Intracellular clearance of ritonavir-boosted Atazanavir | 18 months
  The steady state intracellular CL of ATV/r when administered in adjusted (PBPK model-predicted) doses (300/100mg twice daily) concurrently with standard dose of RIF (600mg) in HIV infected individuals.

SECONDARY OUTCOMES:
Plasma Cmax of ritonavir-boosted Atazanavir when given with 1200mg rifampicin | 18 months
  To evaluate the steady state Cmax of ATV/r, when administered in adjusted doses of 300/100mg b.i.d concurrently with double dose of RIF (1200 mg once daily) in HIV infected individuals.
Plasma AUC of ritonavir-boosted Atazanavir when given with 1200mg rifampicin | 18 months
  To evaluate the steady state AUC of ATV/r, when administered in adjusted doses of 300/100mg b.i.d concurrently with double dose of RIF (1200 mg once daily) in HIV infected individuals.
Plasma Clearance of ritonavir-boosted Atazanavir when given with 1200mg rifampicin | 18 months
  To evaluate the steady state CL of ATV/r, when administered in adjusted doses of 300/100mg b.i.d concurrently with double dose of RIF (1200 mg once daily) in HIV infected individuals.
Intracellular concentration of ritonavir-boosted atazanavir | 18 months
  To evaluate the intracellular PK of ATV/r when administered at standard and at adjusted doses of ATV/r (300/100mg q.d and 300/100mg b.i.d) and RIF (600mg and 1200mg q.d)
Intracellular concentration of DTG | 18 months
  To evaluate the intracellular PK of DTG when administered at standard and at adjusted doses of ATV/r (300/100mg q.d and 300/100mg b.i.d) and RIF (600mg and 1200mg q.d)
Intracellular concentration of RIF | 18 months
  To evaluate the intracellular PK of RIF when administered at standard and at adjusted doses of ATV/r (300/100mg q.d and 300/100mg b.i.d) and RIF (600mg and 1200mg q.d)
Grade 3 adverse events (by DAIDS) | 18 months
  To evaluate the proportion of participants with grade > 3 adverse events by week 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Joint Clinical Research Centre, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
To be finalised, but data management plan is consistent with European law as per EDCTP guidelines.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Will become available after publication of primary endpoint
Access Criteria: To be determined. Website for the consortium is via the URL, with data sharing section not yet developed.
URL: http://pmxafrica.org/Uganda

REFERENCES:
- [Derived] Gausi K, Mugerwa H, Siccardi M, Montanha MC, Lamorde M, Wiesner L, D'Avolio A, McIlleron H, Wilkins E, De Nicolo A, Maartens G, Khoo S, Kityo C, Denti P, Waitt C. Pharmacokinetics and Safety of Twice-daily Ritonavir-boosted Atazanavir With Rifampicin. Clin Infect Dis. 2024 May 15;78(5):1246-1255. doi: 10.1093/cid/ciad700. PMID 37982585
- [Derived] Urbaniak A, Thummel KE, Alade AN, Rettie AE, Prasad B, De Nicolo A, Martin JH, Sheppard DN, Jarvis MF. Experimental pharmacology in precision medicine. Pharmacol Res Perspect. 2023 Dec;11(6):e01147. doi: 10.1002/prp2.1147. No abstract available. PMID 37885364